CLINICAL TRIAL: NCT05432908
Title: Effect of Orofacial Myofunctional Therapy on Unintentional Air Leak From the Oral Cavity in Patients With Obstructive Sleep Apnea Treated With Continuous Positive Upper Airway Pressure (CPAP)
Brief Title: Effect of Orofacial Myofunctional Therapy on Mouth Air Leak in Patients With Sleep Apnea Treated With CPAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties to recruit due to COVID pandemic
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Geraldo Lorenzi Filho, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4525/17/025
Record Dates: First submitted 2022-05-03; First posted 2022-06-27 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: OSA; Apnea+Hypopnea
Keywords: Orofacial Myofunctional Therapy; Oropharyngeal exercises; CPAP; Nasal mask; Air leak; Sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orofacial exercises and oropharyngeal functions (Experimental): Orofacial exercises and oropharyngeal functions.
  Interventions: Behavioral: Orofacial exercises and oropharyngeal functions

INTERVENTIONS:
Behavioral: Orofacial exercises and oropharyngeal functions — Oropharyngeal exercises (derived from speech-language pathology) to the tongue and facial muscles exercises as well stomatognathic functions.

SUMMARY:
To verify the effect of orofacial myofunctional therapy in patients with OSA during the use of CPAP with a nasal mask, on the frequency and leak flow. In addition, the impact on mouth opening frequency, sleep quality, perception of excessive daytime sleepiness, and CPAP adherence will be evaluated.

DETAILED DESCRIPTION:
The use of continuous positive airway pressure (CPAP) with a nasal mask during sleep is the gold standard treatment for moderate to severe obstructive sleep apnea (OSA). However, low adherence to CPAP is the main limiting factor in clinical practice. Recent studies suggest that unintentional air leak through the mouth contributes significantly to poor adherence to CPAP. Orofacial myofunctional therapy (OMT) is effective for treating mild to moderate OSA and has not been tested in patients with mouth air leaks. OSA patients using nasal CPAP and mouth air leaks will be recruited and will use the standard CPAP model and nasal mask during the first and last week of the study to record adherence and home leak. Patients will be treated by performing daily (3 times a day) orofacial myofunctional exercises aimed at strengthening the muscles of the oral cavity. Exercises will be supervised weekly for 3 months. All patients will undergo at the beginning and end of treatment: polysomnography with CPAP and nasal mask, speech-language pathology assessment adequated for OSA (scores ranging from 0 to 241, with higher values indicating greater dysfunction), quality of life questionnaire, and nasosinusal symptoms (SNOT -22), sleep quality (Pittsburgh) and sleepiness (Epworth). Polysomnography will include a pneumotachograph (Hans Rudolph) in the CPAP circuit to record flow and a magnetic jaw movement sensor (Brizzy) to record the episodes of mouth opening. The mouth air leak episodes were considered when they exceeded 20% above baseline (intentional leak with the mask fitted and mouth closed at the beginning of the PSG examination with CPAP) for a minimum of 10 seconds. Leaks ending with arousal or full awakening were considered arousal or full awakening associated with mouth air leak. Mouth opening during the leak episodes was determined by the difference between the amplitude at the end of the leak and the amplitude during the leak. Our hypothesis is that the orofacial myofunctional therapy will reduce mouth leakage in OSA patients treated with CPAP and nasal mask.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosis of OSA (AHI>15 events/h) on use of CPAP (>3 months) with suspect mouth leak as observed by the complaint of morning dry mouth and or CPAP report indicating an excessive air leak

Exclusion Criteria:

* Central Sleep Apnea, oxygen dependent, COPD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Effect of Orofacial Myofunctional Therapy on mouth air leak | 3 months
  The reduction of mouth air leak (L/min) in PSG recordings post Orofacial Myofunctional Therapy

SECONDARY OUTCOMES:
Effect of Orofacial Myofunctional Therapy on the leak in CPAP report | 3 months
  Effect of Orofacial Myofunctional Therapy on the mean value of leak in liters per minute in the CPAP report
Effect of Orofacial Myofunctional Therapy on the adherence to CPAP | 3 months
  Effect of Orofacial Myofunctional Therapy on the mean value of hours of use in the CPAP report
Effect of Orofacial Myofunctional Therapy on the Pittsburgh Sleep Quality Index score | 3 months
  The reduction in questionnaire scores on Pittsburgh Sleep Quality Index, ranging from 0 to 21 (referred to as the global score), with the higher total score indicating worse sleep quality, post-Orofacial Myofunctional Therapy
Effect of Orofacial Myofunctional Therapy on the Epworth Sleepiness Scale score | 3 months
  The reduction in questionnaire scores on the perception of excessive daytime somnolence (Epworth Sleepiness Scale, score ranging from 0 to 24, with a total score ≥10 representing excessive daytime sleepiness) post-Orofacial Myofunctional Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Geraldo Lorenzi-Filho, PhD, Principal Investigator — Hospital das Clínicas HCFMUSP
Locations (1):
- Fundação Zerbini - Instituto do Coração (InCor), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebret M, Martinot JB, Arnol N, Zerillo D, Tamisier R, Pepin JL, Borel JC. Factors Contributing to Unintentional Leak During CPAP Treatment: A Systematic Review. Chest. 2017 Mar;151(3):707-719. doi: 10.1016/j.chest.2016.11.049. Epub 2016 Dec 14. PMID 27986462
- [Background] Camacho M, Certal V, Abdullatif J, Zaghi S, Ruoff CM, Capasso R, Kushida CA. Myofunctional Therapy to Treat Obstructive Sleep Apnea: A Systematic Review and Meta-analysis. Sleep. 2015 May 1;38(5):669-75. doi: 10.5665/sleep.4652. PMID 25348130
- [Background] Valentin A, Subramanian S, Quan SF, Berry RB, Parthasarathy S. Air leak is associated with poor adherence to autoPAP therapy. Sleep. 2011 Jun 1;34(6):801-6. doi: 10.5665/SLEEP.1054. PMID 21629369
- [Background] Lebret M, Arnol N, Martinot JB, Lambert L, Tamisier R, Pepin JL, Borel JC. Determinants of Unintentional Leaks During CPAP Treatment in OSA. Chest. 2018 Apr;153(4):834-842. doi: 10.1016/j.chest.2017.08.017. Epub 2017 Aug 26. PMID 28847549
- [Background] Rotty MC, Suehs CM, Mallet JP, Martinez C, Borel JC, Rabec C, Bertelli F, Bourdin A, Molinari N, Jaffuel D. Mask side-effects in long-term CPAP-patients impact adherence and sleepiness: the InterfaceVent real-life study. Respir Res. 2021 Jan 15;22(1):17. doi: 10.1186/s12931-021-01618-x. PMID 33451313